CLINICAL TRIAL: NCT06379958
Title: A Phase 1, Open-label, 4-Part, Drug-Drug Interaction Study to Evaluate the Effects of Inhibition and Induction of CYP3A4 on the Pharmacokinetics of Leramistat, to Assess the Effect of Leramistat on the Pharmacokinetics of Simvastatin, and to Evaluate the Pharmacokinetic Interaction Between Leramistat and Upadacitinib (RINVOQ®) in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction (DDI) Study of Leramistat in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Modern Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IST-05
Record Dates: First submitted 2024-04-08; First posted 2024-04-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Itraconazole; Phenytoin; Simvastatin; upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Itraconazole 200mg (Active Comparator)
  Interventions: Drug: leramistat 40mg; Drug: Itraconazole 200 mg
- Part 2: Phenytoin 100mg (Active Comparator)
  Interventions: Drug: leramistat 40mg; Drug: Phenytoin 100 Mg Oral Capsule
- Part 3: Simvastatin 40mg (Active Comparator)
  Interventions: Drug: leramistat 40mg; Drug: Simvastatin 40mg
- Part 4: Upadacitinib 15 mg (Active Comparator)
  Interventions: Drug: leramistat 40mg; Drug: Upadacitinib 15 MG

INTERVENTIONS:
Drug: leramistat 40mg — Oral capsule
Drug: Itraconazole 200 mg — Oral capsule
  Arms: Part 1: Itraconazole 200mg
Drug: Phenytoin 100 Mg Oral Capsule — Oral capsule
  Arms: Part 2: Phenytoin 100mg
Drug: Simvastatin 40mg — Oral capsule
  Arms: Part 3: Simvastatin 40mg
Drug: Upadacitinib 15 MG — Oral Capsule
  Arms: Part 4: Upadacitinib 15 mg

SUMMARY:
A DDI study consisting of 4 parts conducted as an open label, fixed sequence study in healthy adult subjects.

ELIGIBILITY:
Principal Inclusion Criteria:

Healthy, adult, male or female of non childbearing potential 18 to 55 years of age.

Principal Exclusion Criteria:

History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.

History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
leramistat: Area under the curve - AUC0-t | 8.5 Weeks
leramistat: Area under the curve - AUC0-24h | 8.5 Weeks
leramistat: Area under the curve - AUC0-inf | 8.5 weeks
leramistat: Maximum observed concentration - Cmax | 8.5 weeks
leramistat: Time of the maximum observed concentration - Tmax | 8.5 weeks
leramistat:Elimination rate constant -Kel | 8.5 weeks
leramistat: Half life - t½ | 8.5 weeks
leramistat: Plasma Clearance -CL/F | 8.5 weeks
leramistat: Volume of distribution - Vz/F | 8.5 weeks

SECONDARY OUTCOMES:
Incidence of adverse event. | 8.5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No